CLINICAL TRIAL: NCT06963307
Title: LUMEN-Dx: Novel Epigenetic Mapping in Cell-Free DNA for the Detection of Lung Cancer
Brief Title: Novel Epigenetic Mapping in Cell-Free DNA for the Detection of Lung Cancer
Acronym: LumenDx
Status: Recruiting | Type: Observational
Sponsor: JaxBio Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 101188111; 101188111 (Other Grant/Funding Number: EU)
Record Dates: First submitted 2025-04-30; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: lung cancer; liquid biopsy; cancer diagnostics; follow-up; minimal residual disease; cell-free DNA; epigenetics; DNA methylation; response to therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected and separated to plasma and buffy coat. Cell-free DNA will be extracted from the plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lung cancer patients: lung cancer patients will be recruited at diagnosis. Blood will be taken before surgery / treatment and after surgery / treatment at the indicated time points.
- non-malignant lung disease: Non-malignant lung disease cohort includes patients with chronic lung disease such as COPD, or acute pneumonia, and will serve as a control group to identify lung cancer and distinguish it from other lung diseases.
- Healthy controls: Healthy individuals will serve as a control group.

SUMMARY:
This trial is a multicenter, open-label, non-interventional controlled study to identify and characterize epigenetic signatures of lung cancer. The goal of this study is to develop a simple blood test that can detect lung cancer with high sensitivity, and assist in the early diagnosis and management of lung cancer.

In particular, the ability to assist existing methods in cancer diagnostics, predict response to treatment, and assess the success of treatment during and after treatment will be examined. In addition, the ability to assess minimal residual disease (MRD) will be evaluated, by taking blood after surgery to remove a tumor or after treatment, and testing whether there is any residual DNA from the tumor using the markers that are found.

The collection of patients and data will be conducted over a period of about a year and a half, with the aim of reaching approximately 300 participants, including patients with lung cancer before and after treatment/surgery and control groups.

DETAILED DESCRIPTION:
During cell death, which occurs frequently in cancerous tissue, DNA from the dead cells is released into the blood. This DNA has a unique epigenetic pattern that can indicate the tissue of origin from which it was released. Therefore, cell-free DNA may serve as a biomarker for monitoring tissues in which there is increased cell death and allow for early detection of disease before it is even visible by other existing methods. In addition, because the epigenetic pattern is dynamic and changes depending on the existing condition, epigenetic changes may allow the identification of the type of disease or serve as a marker for responsiveness to treatment.

The aim of the proposed study is to perform epigenetic mapping in cell-free DNA to identify genomic regions that differ in their epigenetic pattern between lung cancer patients of all histological types, patients with chronic lung diseases, patients with acute pneumonia, and healthy individuals. In particular, the ability to assist existing methods in cancer diagnostics, predict response to treatment, and assess the success of treatment during and after treatment will be examined. In addition, the ability to assess minimal residual disease (MRD) will be examined by taking blood after surgery to remove a tumor or after treatment and testing whether there is any residual DNA from the tumor using the markers that are found. This method may allow early identification of MRD in lung cancer by cell-free DNA in the blood, thus influencing the method of treatment and significantly increasing the chances of survival for patients.

Subjects will be screened for eligibility and then, after signing an Informed Consent Form, the first peripheral blood sample will be obtained.

Lung cancer patients undergoing treatment will donate blood at the following time points: before starting their first systemic treatment (immunotherapy/chemo-immunotherapy) treatment, 4-12 weeks after treatment initiation, and 6-12 months post-treatment.

Lung cancer patients undergoing surgery to remove lung cancer will donate blood at the following time points: before the surgery, 4-6 weeks after surgery, and 6-12 months post-surgery.

Patients with positive or inconclusive low-dose CT findings and negative biopsy results for lung cancer will be recruited to evaluate the ability of the test to assist in a more accurate diagnosis.

Patients with chronic lung disease or acute pneumonia, with no lung cancer diagnosis and 50 healthy volunteers will be recruited as control groups. These participate will donate blood once during the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* Patients diagnosed with lung cancer before systemic therapy.
* Patients with inconclusive LDCT findings.
* Healthy volunteers.
* Patients with chronic lung diseases (COPD, pulmonary emphysema, acute pneumonia).

Exclusion Criteria:

* Subjects who did not sign a consent form.
* Patients with cancer other than lung cancer.
* Patients with HIV or hepatitis.
* Patients with active autoimmune diseases (except lung-localized diseases).
* Pregnant women or individuals unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * 100 patients with various types of lung cancer before starting their first systemic treatment (immunotherapy/chemo-immunotherapy). Samples will be taken before treatment, 4-12 weeks after treatment initiation, and 6-12 months post-treatment.
  * 50 patients undergoing lung cancer surgery. Samples will be collected before surgery, 4-6 weeks after surgery, and 6-12 months post-surgery.
  * 50 patients with positive or inconclusive LDCT findings and negative biopsy results for lung cancer.
  * 50 patients with chronic lung disease or acute pneumonia, with no lung cancer diagnosis.
  * 50 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Define a set of differential epigenetic biomarkers that uniquely identify lung cancer | 12 months from the first blood draw
  Define a set of differential epigenetic biomarkers that uniquely identify lung cancer and can assist in companion diagnostics, evaluate treatment response, predict response to therapy, and detect minimal residual disease following surgery or treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No